CLINICAL TRIAL: NCT01826487
Title: A Phase 3 Efficacy and Safety Study of Ataluren in Patients With Nonsense Mutation Dystrophinopathy
Brief Title: Phase 3 Study of Ataluren in Participants With Nonsense Mutation Duchenne Muscular Dystrophy (nmDMD)
Acronym: ACT DMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTC124-GD-020-DMD; 2012-004527-20 (EudraCT Number)
Record Dates: First submitted 2013-03-26; First posted 2013-04-08 (Estimated); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Muscular Dystrophy, Duchenne; Muscular Dystrophies; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, X-Linked; Genetic Diseases, Inborn
Keywords: Duchenne muscular dystrophy; Dystrophinopathy; Nonsense mutation; Premature stop codon; Becker muscular dystrophy; DMD/BMD; PTC124; Ataluren
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, X-Linked; Genetic Diseases, Inborn | interventions — ataluren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive placebo matching to ataluren orally 3 times a day (TID) at morning, midday, and evening for 48 weeks.
  Interventions: Drug: Placebo
- Ataluren (Experimental): Participants will receive ataluren suspension orally TID, 10 milligrams/kilogram (mg/kg) at morning, 10 mg/kg at midday, and 20 mg/kg at evening (total daily dose 40 mg/kg) for 48 weeks.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be administered as per the dose and schedule specified in the arm.
  Other Names: PTC124
  Arms: Ataluren
Drug: Placebo — Placebo will be administered as per the schedule specified in the arm.
  Arms: Placebo

SUMMARY:
Dystrophinopathy is a disease continuum that includes Duchenne muscular dystrophy, which develops in boys. It is caused by a mutation in the gene for dystrophin, a protein that is important for maintaining normal muscle structure and function. Loss of dystrophin causes muscle fragility that leads to weakness and loss of walking ability. A specific type of mutation, called a nonsense (premature stop codon) mutation is the cause of dystrophinopathy in approximately 10-15 percent (%) of boys with the disease. Ataluren is an orally delivered, investigational drug that has the potential to overcome the effects of the nonsense mutation. The main goal of this Phase 3 study is to evaluate the effect of ataluren on walking ability. The effect of ataluren on physical function, quality of life, and activities of daily living will be evaluated. This study will also provide additional information on the long-term safety of ataluren.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study to determine the efficacy and safety of ataluren in participants with nmDMD.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent (parental/guardian consent if applicable)/assent per local requirements.
* Phenotypic evidence of dystrophinopathy based on the onset of characteristic clinical symptoms or signs (for example; proximal muscle weakness, waddling gait, and Gowers' maneuver) by 6 years of age, an elevated serum creatinine kinase level, and ongoing difficulty with walking.
* Documentation of the presence of a nonsense point mutation in the dystrophin gene as determined by gene sequencing from a laboratory certified by the College of American Pathologists (CAP), the Clinical Laboratory Improvement Act/Amendment (CLIA) or an equivalent organization.
* Documentation that a blood sample has been drawn for confirmation of the presence of a nonsense mutation in the dystrophin gene.
* Use of systemic corticosteroids (prednisone, prednisolone, or deflazacort) for a minimum of 6 months immediately prior to start of study treatment, with no significant change in dosage or dosing regimen (not related to body weight change) for a minimum of 3 months immediately prior to start of study treatment and a reasonable expectation that dosage and dosing regimen will not change significantly for the duration of the study.
* Valid Screening 6-minute walk distance (6MWD) greater than or equal to (≥) 150 meters. Valid Screening 6MWD must have been less than or equal to (≤) 80% of predicted for age and height.
* Results of the 2 Baseline 6MWD results must be determined as valid and results of the Day 2 Baseline 6MWD must be within 20% of the Day 1 Baseline 6MWD.
* Baseline 6MWD (mean of valid Day 1 and Day 2 values) must be no more than a 20% change from the valid Screening 6MWD.
* Confirmed screening laboratory values within the central laboratory ranges (hepatic, renal, and serum electrolyte parameters).
* Willingness to abstain from sexual intercourse or employ an approved method of contraception during the period of study drug administration and 6-week follow-up period.
* Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, laboratory tests, and study restrictions.

Exclusion Criteria:

* Treatment with systemic aminoglycoside antibiotics within 3 months prior to start of study treatment.
* Initiation of systemic corticosteroids therapy within 6 months prior to start of study treatment.
* Change in systemic corticosteroid therapy (for example; change in type of drug, dose modification not related to body weight change, schedule modification, interruption, or reinitiation) within 3 months prior to start of study treatment.
* Any change (initiation, change in type of drug, dose modification, schedule modification,interruption, discontinuation, or reinitiation) in prophylaxis/treatment for congestive heart failure (CHF) within 3 months prior to start of study treatment.
* Ongoing use of coumarin-based anticoagulants (for example; warfarin), phenytoin, tolbutamide, or paclitaxel.
* Prior therapy with ataluren.
* Known hypersensitivity to any of the ingredients or excipients of the study drug.
* Exposure to another investigational drug within 3 months prior to start of study treatment.
* History of major surgical procedure within 6 weeks prior to start of study treatment.
* Ongoing immunosuppressive therapy (other than corticosteroids).
* Ongoing participation in any clinical trial (except for studies specifically approved by PTC Therapeutics).
* Expectation of major surgical procedure (for example; scoliosis surgery) during the 12-month treatment period of the study.
* Requirement for daytime ventilator assistance.
* Uncontrolled clinical symptoms and signs of CHF (American College of Cardiology/American Heart Association Stage C or Stage D).
* Prior or ongoing medical condition (for example; concomitant illness, psychiatric condition, behavioral disorder, alcoholism, drug abuse), medical history, physical findings (for example; lower limb injury that may affect 6MWT performance), electrocardiogram (ECG) findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.

Ages: 7 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2013-03-26 (Actual); Primary Completion 2015-08-20 (Actual); Study Completion 2015-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Spiegel, M.D., Study Director — PTC Therapeutics
Locations (55):
- United States (21):
  - University of California, Los Angeles, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Children's Hospital Colorado - Center for Cancer and Blood Disorders, Aurora, Colorado
  - Child Neurology Center of Northwest Florida, Gulf Breeze, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, Division of Endocrinology, Metabolism and Lipid Research, St Louis, Missouri
  - Columbia University College of Physicians & Surgeons, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Childrens Medical Center Dallas, Texas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital - Childhood Cancer and Blood Disorders, Seattle, Washington
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - The Royal Children's Hospital, Parkville, Victoria
- UZ Leuven, Leuven, Belgium
- Brazil (2):
  - Universidade Federal do Rio de Janeiro - Instituto de Puericultura e Pediatria Martagao Gesteira, Rio de Janeiro
  - Sao Paulo University -HC/FMUSP, São Paulo
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Children's Hospital of Western Ontario, London, Ontario
- Chile (2):
  - Hospital Luis Calvo Mackenna, Santiago, Santiago Metropolitan
  - Hospital Clinico Universidad Catolica, Santiago
- Czechia (2):
  - University Hospital Brno, Brno
  - Motol University Hospital, Prague
- France (4):
  - Hospital de la Timone, Marseille
  - CHU de Nantes, Nantes
  - Hopital Necker - Enfants Malades, Paris
  - Groupe Hospitalier La Pitie-Salpetriere, Paris
- Germany (2):
  - University of Essen-Duisburg, Essen
  - University Hospital Medical Center Freiburg, Freiburg im Breisgau
- Hadassah University Hospital, Jerusalem, Israel
- Italy (4):
  - Policlinico Universitario G. Martino, Messina, Sicily
  - Fondazione IRCS Ca Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Bambino Gesu Hospital, Rome
  - U.O. Complessa di Neuropsichiatria Infantile, Rome
- Medical University of Warsaw, Warsaw, Poland
- Seoul National University Hospital, Seoul, South Korea
- Spain (2):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitari i Politecnic la Fe, Valencia
- Sweden (2):
  - Queen Silvia Children's Hospital, Gothenburg
  - Astrid Lindgren Childrens Hospital, Stockholm
- CHUV Lausanne, Lausanne, Switzerland
- Hacettepe Childrens Hospital, Ankara, Turkey (Türkiye)
- United Kingdom (3):
  - University College London Institute of Child Health, London
  - Royal Manchester Children's Hospital, Manchester
  - The Newcastle upon Tyne Hospitals, NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shieh PB, Elfring G, Trifillis P, Santos C, Peltz SW, Parsons JA, Apkon S, Darras BT, Campbell C, McDonald CM; Members of the Ataluren Phase IIb Study Group; Members of the Ataluren Phase IIb Study Clinical Evaluator Training Group; Members of the ACT DMD Study Group; Members of the ACT DMD Clinical Evaluator Training Group. Meta-analyses of deflazacort versus prednisone/prednisolone in patients with nonsense mutation Duchenne muscular dystrophy. J Comp Eff Res. 2021 Dec;10(18):1337-1347. doi: 10.2217/cer-2021-0018. Epub 2021 Oct 25. PMID 34693725
- [Derived] McDonald CM, Wei LJ, Flanigan KM, Elfring G, Trifillis P, Muntoni F; ACT DMD Clinical Evaluator Training Group; ACT DMD Study Group. Evaluating longitudinal therapy effects via the North Star Ambulatory Assessment. Muscle Nerve. 2021 Nov;64(5):614-619. doi: 10.1002/mus.27396. Epub 2021 Sep 2. PMID 34383312
- [Derived] Campbell C, Barohn RJ, Bertini E, Chabrol B, Comi GP, Darras BT, Finkel RS, Flanigan KM, Goemans N, Iannaccone ST, Jones KJ, Kirschner J, Mah JK, Mathews KD, McDonald CM, Mercuri E, Nevo Y, Pereon Y, Renfroe JB, Ryan MM, Sampson JB, Schara U, Sejersen T, Selby K, Tulinius M, Vilchez JJ, Voit T, Wei LJ, Wong BL, Elfring G, Souza M, McIntosh J, Trifillis P, Peltz SW, Muntoni F; PTC124-GD-007-DMD Study Group; ACT DMD Study Group; Clinical Evaluator Training Groups. Meta-analyses of ataluren randomized controlled trials in nonsense mutation Duchenne muscular dystrophy. J Comp Eff Res. 2020 Oct;9(14):973-984. doi: 10.2217/cer-2020-0095. Epub 2020 Aug 27. PMID 32851872
- [Derived] McDonald CM, Campbell C, Torricelli RE, Finkel RS, Flanigan KM, Goemans N, Heydemann P, Kaminska A, Kirschner J, Muntoni F, Osorio AN, Schara U, Sejersen T, Shieh PB, Sweeney HL, Topaloglu H, Tulinius M, Vilchez JJ, Voit T, Wong B, Elfring G, Kroger H, Luo X, McIntosh J, Ong T, Riebling P, Souza M, Spiegel RJ, Peltz SW, Mercuri E; Clinical Evaluator Training Group; ACT DMD Study Group. Ataluren in patients with nonsense mutation Duchenne muscular dystrophy (ACT DMD): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Sep 23;390(10101):1489-1498. doi: 10.1016/S0140-6736(17)31611-2. Epub 2017 Jul 17. PMID 28728956
- See also: Related Info — http://www.ptcbio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 291 participants were screened for eligibility, of which 61 participants did not meet entry criteria.
Pre-assignment Details: A total of 230 eligible participants were randomized in 1:1 ratio to receive either placebo or ataluren. 2 participants, 1 in each treatment arm, were excluded from intent-to-treat (ITT) population; as they did not have at least 1 valid post-baseline 6-minute walk distance (6MWD) value, a requirement for inclusion in ITT population.
Groups:
- Placebo: Participants received placebo matched to ataluren orally 3 times a day (TID) at morning, midday, and evening for 48 weeks.
- Ataluren: Participants received ataluren suspension orally TID, 10 milligrams/kilogram (mg/kg) at morning, 10 mg/kg at midday, and 20 mg/kg at evening (total daily dose 40 mg/kg) for 48 weeks.
Period: Overall Study
Arm/Group | Placebo | Ataluren
Started | 115 | 115
As-treated Population (All Randomized participants who received any study treatment.) | 115 | 115
ITT Population (Received any study treatment; had a valid baseline, and at least 1 valid post-baseline 6MWD value.) | 114 | 114
Completed | 111 | 110
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: As-treated population included all randomized participants who actually received any study treatment.
Groups:
- Placebo: Participants received placebo matched to ataluren orally TID at morning, midday, and evening for 48 weeks.
- Ataluren: Participants received ataluren suspension orally TID, 10 mg/kg at morning, 10 mg/kg at midday, and 20 mg/kg at evening (total daily dose 40 mg/kg) for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ataluren | Total
Number analyzed (Participants) | 115 | 115 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (1.65) | 8.9 (1.79) | 8.9 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 115 | 115 | 230
6 Minute Walk Distance (6MWD) [Mean (Standard Deviation); unit: meters] — The 6-minute walk distance (6MWD) test is a non-encouraged test performed in a 30 meters long flat corridor, where the participant is instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. Ambulation was assessed via the 6MWD test following standardized procedures by measuring the 6MWD in meters. Participants were not permitted to use assistive devices (walker, long leg braces, or short leg braces) during the 6MWD test.
  meters | 362.69 (81.424) | 364.04 (73.342) | 363.36 (77.322)
Time to Walk/Run 10 Meters [Mean (Standard Deviation); unit: seconds] | 6.83 (2.924) | 6.66 (3.078) | 6.75 (2.996)
Time to Climb 4 Stairs [Mean (Standard Deviation); unit: seconds] — Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  seconds
    number analyzed (Participants) | 112 | 112 | 224
    (all) | 6.76 (7.287) | 5.99 (5.347) | 6.38 (6.389)
Time to Descend 4 Stairs [Mean (Standard Deviation); unit: seconds] — Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  seconds
    number analyzed (Participants) | 109 | 112 | 221
    (all) | 5.05 (5.362) | 5.07 (5.157) | 5.06 (5.247)
Physical Function Total Score as Measured by North Star Ambulatory Assessment (NSAA) [Mean (Standard Deviation); unit: units on a scale] — NSAA comprised tests of 17 abilities, such as ability to stand, rise from floor, get from lying to sitting, get from sitting to standing, raise one's head, stand on one's heels, hop, jump, and run. For each activity, a score of 0, 1, or 2 was recorded, with 0 = "unable to achieve independently," 1 = "modified method but achieves goal independent of physical assistance from another," or 2 = "normal- achieves goal without any assistance." Sum of these 17 scores was reported as ordinal total score, which can be transformed to a linear total score from 0 (worst) to 100 (best). Population: Intent-to-treat (ITT) population included all participants who were randomized and received any study treatment; and had a valid baseline, and at least one valid post-baseline 6MWD value.
  units on a scale
    number analyzed (Participants) | 114 | 114 | 228
    (all) | 60.2 (18.37) | 60.9 (17.97) | 60.6 (18.14)
Baseline 6MWT [Count of Participants; unit: Participants] — The 6MWD test is a non-encouraged test performed in a 30 meters long flat corridor, where the participant is instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. Ambulation was assessed via the 6MWD test following standardized procedures by measuring the 6MWD in meters. Participants were not permitted to use assistive devices (walker, long leg braces, or short leg braces) during the 6MWD test.
  Participants
    <300 meters | 22 | 25 | 47
    >=300 to <400 meters | 52 | 47 | 99
    >=400 meters | 41 | 43 | 84
Pediatric Outcomes Data Collection Instrument (PODCI) Scores [Mean (Standard Deviation); unit: units on a scale] — PODCI includes a Global Functioning Scale and 5 core scales: Upper Extremity & Physical Function,Transfer/Basic Mobility, Sports/Physical Functioning, Pain/Comfort,and Happiness. Following PODCI domains were prespecified in protocol for analysis:Transfers/Basic Mobility domain assesses difficulty experienced in performing routine motor activities in daily life. Sports/Physical Functioning domain assesses difficulty encountered in participating in more active recreational activities. Each domain was scored from 0 (poor outcome/worse health) to 100(the highest level of functioning & least pain). Population: ITT population included all participants who were randomized and received any study treatment; and had a valid baseline, and at least one valid post-baseline 6MWD value.
  units on a scale
    Transfers/Basic Mobility Score: number analyzed (Participants) | 114 | 114 | 228
    Transfers/Basic Mobility Score | 81.4 (15.79) | 83.9 (13.10) | 82.7 (14.53)
    Sports/Physical Functioning Score: number analyzed (Participants) | 114 | 114 | 228
    Sports/Physical Functioning Score | 56.0 (20.94) | 56.2 (18.94) | 56.1 (19.92)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 6MWD at Week 48
Description: The 6MWD test is a non-encouraged test performed in a 30 meters long flat corridor, where the participant is instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. Ambulation was assessed via the 6MWD test following standardized procedures by measuring the 6MWD in meters. Participants were not permitted to use assistive devices (walker, long leg braces, or short leg braces) during the 6MWD test. Participants with confirmed loss of ambulation at a particular visit were assigned a 6MWD result of 0. Baseline and Week 48 6MWD values are each the average of two valid 6MWD values, or a single available value if one was missing.
Time Frame: Baseline, Week 48
Population: ITT population included all participants who were randomized and received any study treatment; and had a valid baseline, and at least one valid post-baseline 6MWD value. Multiple imputation was applied to impute missing values within the treatment groups.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Placebo | Ataluren
Number analyzed (Participants) | 114 | 114
meters | -60.67 (9.323) | -47.69 (9.247)
Statistical Analysis 1: Comparison: Placebo vs Ataluren; Analysis was performed using analysis of covariance (ANCOVA) method including stratification factors for age (less than [<] 9 years versus [vs.] greater than or equal to [>=] 9 years), duration of use of corticosteroids at baseline (approx. >=6 to <12 months vs. >=12 months), and baseline 6MWD category (>=350 meters vs <350 meters), as well as baseline 6MWD as covariate; Test type: Other; p = 0.213, Mixed Models Analysis — Threshold for significance at 0.05. Secondary endpoints were tested for significance, only if the primary endpoint was statistically significant; Mean Difference (Final Values) = 12.98, 95% CI 2-sided [-7.44 to 33.39], Standard Error of Mean 10.415

2. Secondary Outcome: Time to 10 Percent (%) Persistent Worsening in 6MWD
Description: The 6MWD test is a non-encouraged test performed in a 30 meters long flat corridor, where the participant is instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. Ambulation was assessed via the 6MWD test following standardized procedures by measuring the 6MWD in meters. Participants were not permitted to use assistive devices (walker, long leg braces, or short leg braces) during the 6MWD test. Time to 10% persistent worsening in 6MWD was defined as the last time that 6MWD was not 10% worse compared with baseline. Time to 10% persistent worsening in 6MWD <300 meters, >=300 to 400 meters, and >=400 meters was evaluated. For participants who did not have 10% 6MWD worsening or who were removed from study, time to 10% 6MWD worsening was censored at the time of the last 6MWD test. Participants who became non-ambulatory were considered to have 10% worsening.
Time Frame: Baseline to Week 48
Population: ITT population included all participants who were randomized and received any study treatment; and had a valid baseline, and at least one valid post-baseline 6MWD value. Multiple imputation was applied to impute missing values within treatment groups. Here, 'Number analyzed 'signifies participants evaluable for specified categories.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Ataluren
Number analyzed (Participants) | 114 | 114
days
  <300 meters: number analyzed (Participants) | 21 | 24
  <300 meters | 56 [1.0 to 111.0] | 164 [1.0 to 225.0]
  >=300 to <400 meters: number analyzed (Participants) | 52 | 47
  >=300 to <400 meters | 280 [169.0 to NA] — Due to smaller number of participants with an event, upper limit of 95% confidence interval (CI) could not be calculated. | NA [280.0 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI could not be calculated.
  >=400 meters: number analyzed (Participants) | 41 | 43
  >=400 meters | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% CI could not be calculated. | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% CI could not be calculated.

3. Secondary Outcome: Change From Baseline in Time to Walk/Run 10 Meters at Week 48
Description: During the test for walking/running 10 meters, the method of walk/run used by the participant was categorized as follows: 1. Unable to walk independently; 2. Unable to walk independently but can walk with support from a person or with assistive device (full leg calipers [knee-ankle-foot orthoses ] or walker); 3. Highly adapted gait, wide-based lordotic gait, cannot increase walking speed; 4. Moderately adapted gait, can pick up speed but cannot run; 5. Able to pick up speed but runs with a double stance phase (that is, cannot achieve both feet off the ground); 6. Runs and gets both feet off the ground (with no double stance phase). If the time taken to perform a test exceeded 30 seconds or if a participant could not perform the test due to disease progression, a value of 30 seconds was used. A cumulative change from baseline data has been reported.
Time Frame: Baseline, Week 48
Population: ITT population included all participants who were randomized and received any study treatment; and had a valid baseline, and at least one valid post-baseline 6MWD value. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Ataluren
Number analyzed (Participants) | 110 | 109
seconds | 3.47 (6.393) | 2.27 (5.216)

4. Secondary Outcome: Change From Baseline in Time to Climb 4 Stairs at Week 48
Description: During the test for stair-climbing, the method of climbing used by the participant was categorized as follows: 1. Unable to up climb 4 standard stairs; 2. Climbs 4 standard stairs "marking time" (climbs one foot at a time, with both feet on a step before moving to next step), using both arms on one or both handrails; 3. Climbs 4 standard stairs "marking time" (climbs one foot at a time, with both feet on a step before moving to next step), using one arm on one handrail; 4. Climbs 4 standard stairs "marking time" (climbs one foot at a time, with both feet on a step before moving to next step), not needing handrail; 5. Climbs 4 standard stairs alternating feet, needs handrail for support; 6. Climbs 4 standard stairs alternating feet, not needing handrail support. A cumulative change from baseline data has been reported.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Ataluren
Number analyzed (Participants) | 103 | 105
seconds | 4.46 (7.310) | 2.65 (5.297)

5. Secondary Outcome: Change From Baseline in Time to Descend 4 Stairs at Week 48
Description: During the test for stair-descending, the method of descending used by the participant was categorized as follows: 1. Unable to descend 4 standard stairs; 2. Descends 4 standard stairs "marking time" (climbs one foot at a time, with both feet on a step before moving to next step), using both arms on one or both handrails; 3. Descends 4 standard stairs "marking time" (climbs one foot at a time, with both feet on a step before moving to next step), using one arm on one handrail; 4. Descends 4 standard stairs "marking time" (climbs one foot at a time, with both feet on a step before moving to next step), not needing handrail; 5. Descends 4 standard stairs alternating feet, needs handrail for support; 6. Descends 4 standard stairs alternating feet, not needing handrail support. A cumulative change from baseline data has been reported.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Ataluren
Number analyzed (Participants) | 100 | 106
seconds | 3.97 (7.854) | 2.15 (5.306)

6. Other Pre Specified Outcome: Change From Baseline in Physical Function Total Score as Measured by NSAA at Week 48
Description: Physical function was assessed via the NSAA, a functional scale specifically designed for ambulant Duchenne muscular dystrophy (DMD) participants. The assessment comprised tests for 17 abilities of a participant, such as ability to stand, rise from the floor, get from lying to sitting, get from sitting to standing, raise one's head, stand on one's heels, hop, jump, and run. For each activity, a score of 0, 1, or 2 was recorded, with 0 = "unable to achieve independently," 1 = "modified method but achieves goal independent of physical assistance from another," or 2 = "normal- achieves goal without any assistance." The sum of these scores (except for 'raise one's head' activity score) was reported as the ordinal total score, which was transformed to a linear total score ranging from 0 (worst) to 100 (best). Participants with confirmed loss of ambulation at a particular visit were assigned a score of 0.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ataluren
Number analyzed (Participants) | 108 | 106
units on a scale | -8.4 (10.65) | -6.3 (10.64)

7. Other Pre Specified Outcome: Number of Participants With Change From Baseline in Activities of Daily Living and Disease Status at Week 48, as Assessed by a Standardized Survey Administered by Site Personnel
Description: Changes in activities of daily living and disease symptoms were captured via a DMD-specific survey administered by Site personnel. At screening or baseline, the participant and/or parent/caregiver were asked to identify any activities of daily living (for example, ambulation, balance, personal hygiene/grooming, dressing and undressing, self-feeding, using the bathroom, handwriting, school performance, behavior or energy level) or symptoms that were affected by the participant's DMD. At post-baseline visit (Week 48), the same participant and/or parent/caregiver was asked to describe any changes from baseline in those activities of daily living/symptoms, within the following categories: physical functioning; general energy level; cognition/school function; emotional/social functioning; and sleep. Changes from baseline were reported on a 5-point Likert scale: 1 (much worse), 2 (slightly worse), 3 (unchanged), 4 (slightly better), or 5 (much better).
Time Frame: Baseline, Week 48
Population: ITT population included all participants who were randomized and received any study treatment; and had a valid baseline, and at least one valid post-baseline 6MWD value. Here, 'Number analyzed 'signifies participants evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ataluren
Number analyzed (Participants) | 114 | 114
Participants
  Physical Functioning: Upper Extremity Activity: number analyzed (Participants) | 82 | 88
  Physical Functioning: Upper Extremity Activity: Much better | 1 | 4
  Physical Functioning: Upper Extremity Activity: Slightly better | 7 | 7
  Physical Functioning: Upper Extremity Activity: Unchanged | 67 | 73
  Physical Functioning: Upper Extremity Activity: Slightly worse | 6 | 2
  Physical Functioning: Upper Extremity Activity: Much worse | 1 | 2
  Physical Functioning: Walking: number analyzed (Participants) | 112 | 108
  Physical Functioning: Walking: Much better | 5 | 8
  Physical Functioning: Walking: Slightly better | 13 | 16
  Physical Functioning: Walking: Unchanged | 57 | 60
  Physical Functioning: Walking: Slightly worse | 19 | 21
  Physical Functioning: Walking: Much worse | 18 | 3
  Physical Functioning: Climbing Stairs: number analyzed (Participants) | 105 | 110
  Physical Functioning: Climbing Stairs: Much better | 4 | 4
  Physical Functioning: Climbing Stairs: Slightly better | 8 | 13
  Physical Functioning: Climbing Stairs: Unchanged | 61 | 65
  Physical Functioning: Climbing Stairs: Slightly worse | 17 | 15
  Physical Functioning: Climbing Stairs: Much worse | 15 | 13
  Physical Functioning: Other: number analyzed (Participants) | 65 | 68
  Physical Functioning: Other: Much better | 4 | 5
  Physical Functioning: Other: Slightly better | 9 | 10
  Physical Functioning: Other: Unchanged | 38 | 44
  Physical Functioning: Other: Slightly worse | 7 | 8
  Physical Functioning: Other: Much worse | 7 | 1
  Cognition/Social Functioning: number analyzed (Participants) | 92 | 104
  Cognition/Social Functioning: Much better | 6 | 5
  Cognition/Social Functioning: Slightly better | 12 | 20
  Cognition/Social Functioning: Unchanged | 71 | 74
  Cognition/Social Functioning: Slightly worse | 3 | 3
  Cognition/Social Functioning: Much worse | 0 | 2
  Emotional/Social Functioning: number analyzed (Participants) | 94 | 105
  Emotional/Social Functioning: Much better | 3 | 8
  Emotional/Social Functioning: Slightly better | 9 | 21
  Emotional/Social Functioning: Unchanged | 75 | 68
  Emotional/Social Functioning: Slightly worse | 5 | 6
  Emotional/Social Functioning: Much worse | 2 | 2
  General Energy Level: number analyzed (Participants) | 83 | 89
  General Energy Level: Much better | 3 | 8
  General Energy Level: Slightly better | 12 | 12
  General Energy Level: Unchanged | 54 | 63
  General Energy Level: Slightly worse | 11 | 5
  General Energy Level: Much worse | 3 | 1
  Sleep: number analyzed (Participants) | 85 | 91
  Sleep: Much better | 3 | 3
  Sleep: Slightly better | 4 | 8
  Sleep: Unchanged | 73 | 76
  Sleep: Slightly worse | 5 | 2
  Sleep: Much worse | 0 | 2
  Other: number analyzed (Participants) | 23 | 23
  Other: Much better | 0 | 1
  Other: Slightly better | 5 | 6
  Other: Unchanged | 15 | 13
  Other: Slightly worse | 2 | 3
  Other: Much worse | 1 | 0

8. Other Pre Specified Outcome: Change From Baseline in PODCI Transfers/Basic Mobility and Sports/Physical Functioning Scores at Week 48
Description: Changes in health-related quality of life (HRQL) were measured via the PODCI questionnaire that has been shown to correlate with disease progression and clinical outcome measures in DMD. PODCI includes a Global Functioning Scale and 5 core scales: Upper Extremity and Physical Function,Transfer/Basic Mobility, Sports/Physical Functioning, Pain/Comfort,and Happiness. The following PODCI domains were prespecified in the protocol for analysis:Transfers/Basic Mobility domain assesses difficulty experienced in performing routine motor activities in daily life. Sports/Physical Functioning domain assesses difficulty encountered in participating in more active recreational activities. Each domain was scored from 0 to 100, with 0 representing a poor outcome/worse health, while 100 representing the highest level of functioning and least pain.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ataluren
Number analyzed (Participants) | 110 | 109
units on a scale
  Transfers/Basic Mobility Score | -8.8 (15.80) | -6.6 (14.76)
  Sports/Physical Functioning Score | -7.3 (15.87) | -5.6 (15.91)

9. Other Pre Specified Outcome: Ataluren Plasma Concentration
Description: Plasma samples for the determination of ataluren concentrations were analyzed using a validated high performance liquid chromatography with tandem mass spectrometry (HPLC/MS-MS) method with a lower limit of quantitation of 0.5 micrograms/milliliter (mcg/mL).
Time Frame: Weeks 8, 16, 24, 32, 40, and 48
Population: As-treated population included all randomized participants who actually received any study treatment. Here, 'Number analyzed 'signifies participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Ataluren
Number analyzed (Participants) | 115
mcg/mL
  Week 08: number analyzed (Participants) | 113
  Week 08 | 4.230 (5.3913)
  Week 16: number analyzed (Participants) | 113
  Week 16 | 3.429 (3.9275)
  Week 24: number analyzed (Participants) | 112
  Week 24 | 3.323 (3.6135)
  Week 32: number analyzed (Participants) | 113
  Week 32 | 3.480 (3.1053)
  Week 40: number analyzed (Participants) | 111
  Week 40 | 3.997 (4.7615)
  Week 48: number analyzed (Participants) | 110
  Week 48 | 3.544 (3.8082)

10. Other Pre Specified Outcome: Study Drug Compliance
Description: Study drug compliance was assessed by quantification of used and unused study drug. Compliance was assessed in terms of the percentage of drug actually taken relative to the amount that should have been taken during the study.
Time Frame: Baseline to Week 48
Population: As-treated population included all randomized participants who actually received any study treatment.
Measure: Mean (Standard Deviation); unit: percentage of drug
Arm/Group | Placebo | Ataluren
Number analyzed (Participants) | 115 | 115
percentage of drug | 95.1 (9.43) | 95.7 (7.57)

11. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. Treatment-emergent adverse event (TEAE) was defined as an adverse event that occurred or worsened in the period extending from first dose of study drug to 6 weeks after the last dose of study drug. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline up to Week 54
Population: As-treated population included all randomized participants who actually received any study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ataluren
Number analyzed (Participants) | 115 | 115
percentage of participants | 87.8 | 89.6

ADVERSE EVENTS:
Time Frame: Baseline up to 6 weeks after the last dose of study drug (Week 54)
Description: As-treated population included all randomized participants who actually received any study treatment.
Arm/Group | Placebo | Ataluren
Serious Adverse Events (participants affected / at risk) | 4/115 | 4/115
Other Adverse Events (participants affected / at risk) | 99/115 | 103/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=115) | Ataluren (N=115)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=115) | Ataluren (N=115)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Right ventricular hypertrophy (Cardiac disorders) | 0 | 2
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Myocardial fibrosis (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 4 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Hyperaldosteronism (Endocrine disorders) | 1 | 0
Astigmatism (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 2 | 0
Eye allergy (Eye disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0
Eye movement disorder (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0
Myopia (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 20
Abdominal pain upper (Gastrointestinal disorders) | 13 | 9
Abdominal pain (Gastrointestinal disorders) | 5 | 7
Abdominal discomfort (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 10 | 3
Flatulence (Gastrointestinal disorders) | 1 | 2
Abnormal faeces (Gastrointestinal disorders) | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 21 | 26
Nausea (Gastrointestinal disorders) | 7 | 7
Tooth crowding (Gastrointestinal disorders) | 0 | 2
Malocclusion (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 12 | 16
Disease progression (General disorders) | 14 | 9
Abasia (General disorders) | 0 | 3
Oedema peripheral (General disorders) | 0 | 3
Fatigue (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Influenza like illness (General disorders) | 2 | 1
Gait disturbance (General disorders) | 1 | 0
Malaise (General disorders) | 3 | 0
Thirst (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Allergy to chemicals (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 2 | 2
Rhinitis allergic (Immune system disorders) | 0 | 1
Allergy to vaccine (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 0
Ear infection (Infections and infestations) | 1 | 6
Gastroenteritis (Infections and infestations) | 4 | 5
Influenza (Infections and infestations) | 5 | 3
Bronchitis (Infections and infestations) | 3 | 2
Conjunctivitis infective (Infections and infestations) | 0 | 2
Fungal skin infection (Infections and infestations) | 1 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 2
Gastrointestinal viral infection (Infections and infestations) | 0 | 2
Hordeolum (Infections and infestations) | 3 | 2
Eye infection (Infections and infestations) | 1 | 1
Gingivitis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 4 | 1
Lung infection (Infections and infestations) | 0 | 1
Acute tonsillitis (Infections and infestations) | 1 | 0
Adenoiditis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 2 | 0
Gingival infection (Infections and infestations) | 1 | 0
Helminthic infection (Infections and infestations) | 1 | 0
Infected bites (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 22 | 24
Upper respiratory tract infection (Infections and infestations) | 6 | 11
Rhinitis (Infections and infestations) | 4 | 8
Pharyngitis (Infections and infestations) | 4 | 4
Tonsillitis (Infections and infestations) | 2 | 3
Sinusitis (Infections and infestations) | 2 | 5
Viral infection (Infections and infestations) | 3 | 3
Nail infection (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 2
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 2 | 1
Parasitic gastroenteritis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 1
Mycoplasma infection (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Rubella (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 20 | 21
Contusion (Injury, poisoning and procedural complications) | 4 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 7 | 3
Laceration (Injury, poisoning and procedural complications) | 1 | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 4 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 2
Electrical burn (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0
Renin increased (Investigations) | 3 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 5
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 2
Abnormal weight gain (Metabolism and nutrition disorders) | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0
Hypervitaminosis D (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 3
Growing pains (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 | 0
Lordosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Headache (Nervous system disorders) | 21 | 21
Autism (Nervous system disorders) | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 2
Petit mal epilepsy (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 3
Aggression (Psychiatric disorders) | 0 | 2
Sleep disorder (Psychiatric disorders) | 0 | 2
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Negativism (Psychiatric disorders) | 0 | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Dysphemia (Psychiatric disorders) | 1 | 0
Middle insomnia (Psychiatric disorders) | 1 | 0
Mood swings (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 7
Dysuria (Renal and urinary disorders) | 3 | 2
Enuresis (Renal and urinary disorders) | 1 | 2
Bladder trabeculation (Renal and urinary disorders) | 0 | 1
Flank pain (Renal and urinary disorders) | 0 | 1
Hypercalciuria (Renal and urinary disorders) | 1 | 0
Myoglobinuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 2
Polyuria (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Urine abnormality (Renal and urinary disorders) | 2 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Genital discomfort (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 4
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 0 | 1
Aortic dilatation (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 3 | 0
Haematoma (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.